CLINICAL TRIAL: NCT00036790
Title: An Open-Label Phase I Dose Escalation Trial To Evaluate The Safety And Pharmacokinetics Of Motexafin Gadolinium And Doxorubicin Chemotherapy In The Treatment Of Advanced Malignancies
Brief Title: Motexafin Gadolinium and Doxorubicin in Treating Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000069322; P30CA014520 (NIH); WCCC-CO-01910; PCI-PCYC-0207; NCI-G02-2061
Record Dates: First submitted 2002-05-13; First posted 2003-01-27 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2015-09

CONDITIONS: Breast Cancer; Chronic Myeloproliferative Disorders; Colorectal Cancer; Head and Neck Cancer; Leukemia; Lung Cancer; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic/Myeloproliferative Diseases; Prostate Cancer; Small Intestine Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; isolated plasmacytoma of bone; extramedullary plasmacytoma; refractory multiple myeloma; Waldenstrom macroglobulinemia; stage III multiple myeloma; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; small intestine lymphoma; unspecified adult solid tumor, protocol specific; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; meningeal chronic myelogenous leukemia; untreated adult acute lymphoblastic leukemia; untreated adult acute myeloid leukemia; refractory hairy cell leukemia; chronic myelomonocytic leukemia; T-cell large granular lymphocyte leukemia; acute undifferentiated leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; secondary acute myeloid leukemia; prolymphocytic leukemia; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome; chronic eosinophilic leukemia; chronic neutrophilic leukemia; recurrent non-small cell lung cancer; recurrent small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; extensive stage small cell lung cancer; limited stage small cell lung cancer; recurrent breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; recurrent colon cancer; stage III colon cancer; stage IV colon cancer; recurrent prostate cancer; stage III prostate cancer; stage IV prostate cancer; recurrent lip and oral cavity cancer; stage III lip and oral cavity cancer; stage IV lip and oral cavity cancer; recurrent paranasal sinus and nasal cavity cancer; stage III paranasal sinus and nasal cavity cancer; stage IV paranasal sinus and nasal cavity cancer; recurrent metastatic squamous neck cancer with occult primary; recurrent hypopharyngeal cancer; stage III hypopharyngeal cancer; stage IV hypopharyngeal cancer; recurrent laryngeal cancer; stage III laryngeal cancer; stage IV laryngeal cancer; recurrent oropharyngeal cancer; stage III oropharyngeal cancer; stage IV oropharyngeal cancer; recurrent nasopharyngeal cancer; stage III nasopharyngeal cancer; stage IV nasopharyngeal cancer; atypical chronic myeloid leukemia; myelodysplastic/myeloproliferative disease, unclassifiable; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12)
MeSH Terms: conditions — Breast Neoplasms; Myeloproliferative Disorders; Colorectal Neoplasms; Head and Neck Neoplasms; Leukemia; Lung Neoplasms; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic-Myeloproliferative Diseases; Prostatic Neoplasms; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Waldenstrom Macroglobulinemia; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Hairy Cell; Leukemia, Myelomonocytic, Chronic; Leukemia, Large Granular Lymphocytic; Leukemia, Biphenotypic, Acute; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Prolymphocytic; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Mycosis Fungoides; Sezary Syndrome; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Neutrophilic, Chronic; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Colonic Neoplasms; Mouth Neoplasms; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Oropharyngeal Neoplasms; Nasopharyngeal Neoplasms; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Lymphoma, B-Cell, Marginal Zone; Congenital Abnormalities | interventions — Doxorubicin; motexafin gadolinium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: doxorubicin hydrochloride
Drug: motexafin gadolinium

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Motexafin gadolinium may increase the effectiveness of doxorubicin by making tumor cells more sensitive to the drug.

PURPOSE: Phase I trial to study the effectiveness of combining motexafin gadolinium with doxorubicin in treating patients who have recurrent or metastatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of motexafin gadolinium and doxorubicin in patients with advanced malignancies.
* Determine the dose-limiting toxicity of this regimen in these patients.
* Determine the safety and tolerability of this regimen in these patients.
* Determine the pharmacokinetics of this regimen in these patients.
* Evaluate the tumor response in patients treated with this regimen.

OUTLINE: This is a dose-escalation, multicenter study. Patients are assigned to 1 of 2 groups.

Group A:

* Course 1: Patients receive motexafin gadolinium IV over 30 minutes on days 1, 8, 9, and 10 and doxorubicin IV over 15 minutes on day 8.
* Course 2: 28 days after the beginning of course 1, patients receive doxorubicin IV over 15 minutes.
* Courses 3-6: Beginning 21 days after course 2, patients receive doxorubicin IV over 15 minutes on day 1 and motexafin gadolinium IV over 30 minutes on days 1-3. Treatment repeats every 21 days.

Group B:

* Course 1: Patients receive motexafin gadolinium IV over 30 minutes on day 1 and doxorubicin IV over 15 minutes on day 8.
* Course 2: 28 days after the beginning of course 1, patients receive doxorubicin IV over 15 minutes on day 1 and motexafin gadolinium IV over 30 minutes on days 1-3.
* Courses 3-6: Beginning 21 days after course 2, patients receive doxorubicin and motexafin gadolinium as in group A.

Treatment in both groups continues for up to 6 courses in the absence of disease progression, unacceptable toxicity, or a cumulative doxorubicin dose of 450 mg/m^2.

Cohorts of 3-6 patients receive escalating doses of doxorubicin and motexafin gadolinium until the maximum tolerated dose (MTD) is determined. The MTD is defined as the highest dose at which no more than 0 of 3 or 1 of 6 patients experience dose-limiting toxicity.

Patients are followed at 1 and 2 months.

PROJECTED ACCRUAL: A total of 3-48 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced malignancy that is considered incurable

  * Recurrent or metastatic disease
  * Relapsed solid tumors include, but are not limited to the following sites:

    * Lung
    * Breast
    * Colon
    * Prostate
    * Head and neck
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex

* Not specified

Menopausal status

* Not specified

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* AST and ALT no greater than 2 times upper limit of normal

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* LVEF greater than 45% at rest
* No prior myocardial infarction
* No congestive heart failure
* No clinically significant ventricular arrhythmias

Other:

* No history of HIV infection
* No history of porphyria
* No glucose-6-phosphate dehydrogenase deficiency
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 6 months after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 28 days since prior chemotherapy
* No prior lifetime cumulative doxorubicin exposure of more than 300 mg/m^2
* No other concurrent cytotoxic chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 28 days since prior radiotherapy
* No concurrent radiotherapy

Surgery:

* No concurrent surgery

Other:

* At least 14 days since prior multidrug resistance-modulating drugs (e.g., PSC833 or cyclosporine)
* No other concurrent antineoplastic or investigational agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-02; Primary Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Markus Renschler, MD, Study Chair — Pharmacyclics LLC.
Locations (2):
- United States (2):
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin